CLINICAL TRIAL: NCT03827252
Title: Identification of Respiratory Stability Mechanisms During Skin-to-skin Care in Premature Infants in the Neonatal Intensive Care Unit: Infant-parent Vegetative Functions Coupling
Brief Title: Respiratory Stability and Vegetative Coupling During Neonatal Skin-to-skin Care
Acronym: PO-A-PO-PREMA
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2017_843_0008
Record Dates: First submitted 2019-01-31; First posted 2019-02-01 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Premature Infant
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The main purpose of this study is to identify and to determine the involvement of cardio-respiratory coordination mechanisms during SSC between the preterm infant and his (her) parent.

DETAILED DESCRIPTION:
The skin to skin care (SSC) is a technique that proceeds by laying the neonate ventrally on the parent's chest. Many positive effects are recognized as due to SSC i.e, maintaining the infant's body temperature, better sleep organization, neurocognitive development and cardio-respiratory stability, more strength in parent-infant affective relations, reduction in neonatal and parental stress, more success in feeding with breast milk. Nowadays, SSC is generalized in modern Neonatal Intensive Care Units as part of developmental care. However, the mechanisms involved in SSC are not totally understood. The hypothesis in this study is that the cardio-respiratory stability results partially from the intervention of the coordination between cardiac and respiratory activities. These suppose the involvement of complex mechanisms of cardio-respiratory coordination including neuro-autonomous loops with chemoreceptors and baroreceptors, bulbar vasomotor and respiratory regulatory centers, ortho-parasympathetic neuronal and chemical pathways and cardiac, vascular and lung effectors. In this study the identification of these characteristics will be performed by processing signals of ECG, SaO2 (arterial oxygen saturation), respiratory movements, perfusion index, cutaneous and ambient temperature extracted from the clinical monitoring systems. Each preterm infant included in the study will be explored twice, 5-10 days apart. The explorations will be carried out on 3 steps: before (at least 30 minutes), during (at least 60 minutes) and after (≥ 60 minutes) the SSC session. Each patient will participate in the study for 10 days at maximum. Inclusions in the study will last for a total period of 18 months and 10 days. The cardio-respiratory coordination will be assessed using coordigram technique, corresponding to the proportion of time with > 0.7 amplitude on spectral density.

ELIGIBILITY:
Inclusion Criteria:

* Premature infant from 28weeks + 0 day to 36 weeks + 6 days gestational corrected age
* At least 72 hours postnatal age
* Benefiting skin-to-skin care

Exclusion Criteria:

* Severe congenital malformation and nervous system dysfunction (e.g., Ondine Sd)
* Septic shock
* Mechanical ventilation support
* Severe pulmonary arterial hypertension
* Analgesia morphinics at high dosage and curare

Ages: 28 Weeks to 36 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Premature infant from 28weeks + 0 day to 36 weeks + 6 days gestational corrected age
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2018-09-07 (Actual); Primary Completion 2019-12-11 (Actual); Study Completion 2020-09-12 (Actual)

PRIMARY OUTCOMES:
Cardio-respiratory coordination index | 10 days
  Percentage of time during the recording that fulfills the criteria of coordination ( > 0.7 amplitude of spectra in coordigram)

SECONDARY OUTCOMES:
Cardio-respiratory coordination index by phase analysis technique | 10 days
Correlation between cardio-respiratory coordination index and SaO2 | 10 days
Correlation of temperatures (infant, parent) and cardio-respiratory coordination index | 10 days

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens-Picardie, Amiens, France

IPD SHARING:
Plan to Share IPD: No